CLINICAL TRIAL: NCT01518842
Title: Effect of Intravitreal Bone Marrow Stem Cells on Ischemic Retinopathy
Acronym: RetinaCell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD - Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Siqueira Research Center
Record Dates: First submitted 2012-01-22; First posted 2012-01-26 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Ischemia
Keywords: ischemic retinopathy, stem cell,bone marrow
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: intravitreal injection of autologous bone marrow stem cells
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- test group intravitreal stem cell (Experimental): Open-label study of Ischemic Retinopathy patients with best-corrected visual acuity (BCVA) worse than 20/200.
  Intervention: Biological: intravitreal injection of autologous bone marrow stem cells
  Interventions: Biological: Intravitreal Bone Marrow Stem Cells

INTERVENTIONS:
Biological: Intravitreal Bone Marrow Stem Cells — One intravitreal injection of a 0.1-ml cell suspension containing around 10x106 bone marrow mononuclear stem cells(BMMSC). All treatments were performed by a single retinal specialist using topical proparacaine drops under sterile conditions (eyelid speculum and povidone-iodine). Autologous BMMSC were injected into the vitreous cavity using a 27 gauge needle inserted through the inferotemporal pars plana 3.0 - 3.5 mm posterior to the limbus. After the injection, central retinal artery perfusion was confirmed with indirect ophthalmoscopy. Patients were instructed to instill one drop of 0.3% ciprofloxacin into the injected eye four times daily for 1 week after the procedure.

SUMMARY:
This study aims to evaluate the behavior of the intravitreal use of bone marrow derived stem cells in patients with ischemic retinopathy.

DETAILED DESCRIPTION:
Evaluate the effects on visual acuity, electroretinography, fluorescein angiography and optical coherence tomography in 30 patients with ischemic retinopathy, including diabetic retinopathy with severe loss of retinal capillaries undergoing intravitreal injection of bone marrow derived stem cells.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Ischemic Retinopathy
* Enlargement of foveal avascular zone-FAZ (ischaemia or capillary drop out of >30% on Fluorescein retinography
* logarithm of minimum angle of resolution (logMAR) BCVA of 1.0 (Snellen equivalent, 20/200) or worse
* Able (in the Investigator's opinion) and willing to comply with all study requirements

Exclusion Criteria:

* previous ocular surgery other than cataract
* presence of cataract or other media opacity that would influence ocular fundus documentation and adequate ERG and visual field evaluation
* other ophthalmic disease like glaucoma and uveitis
* previous history of blood disorders like leukemia
* known allergy to fluorescein or indocyanine green

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2018-10 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in size of FAZ at 48 weeks | 1 day to 48 weeks

SECONDARY OUTCOMES:
Change in central foveal thickness and best corrected visual acuity at 48 weeks | 1 day to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD, PhD, Principal Investigator — Rubens Siqueira Research Center
Locations (1):
- Rubens Siqueira Research Center, São José do Rio Preto, São Paulo, Brazil

REFERENCES:
- [Background] Siqueira RC, Messias A, Gurgel VP, Simoes BP, Scott IU, Jorge R. Improvement of ischaemic macular oedema after intravitreal injection of autologous bone marrow-derived haematopoietic stem cells. Acta Ophthalmol. 2015 Mar;93(2):e174-6. doi: 10.1111/aos.12473. Epub 2014 Jun 22. No abstract available. PMID 24954079